CLINICAL TRIAL: NCT01152866
Title: An Observational Study Using Subcutaneous Ovidrel (Choriogonadotrophin Alfa) for Induction of Final Follicular Maturation and Early Luteinisation in Women Undergoing Ovarian Stimulation With Recombinant-human Follicle Stimulating Hormone (r-hFSH [Gonal-F®]).
Brief Title: An Open Label, Canadian Phase IIIb Study With Ovidrel in Ovulation Induction (OI) and Assisted Reproductive Technique (ART)
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Irene Kavanagh/Medical Research Manager, EMD Serono a division of EMD Canada Inc.
Other Study IDs: 24662
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Ovulation Induction; Infertility
Keywords: Multifollicular stimulation; Pregnancy; Reproductive Techniques, Assisted; Fertilization in Vitro; Infertility
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples

INTERVENTIONS:
Drug: Choriogonadotropin alpha (r-hCG) — Choriogonadotropin alpha 250 μg was administered subcutaneously on the day following the last dose of follitropin alpha (Gonal-F).
  Other Names: Ovidrel

SUMMARY:
With the development of the recombinant gonadotrophins, the use of human source proteins for the production of hormones has become unnecessary. These proteins, which are found in urinary preparations, have been thought to cause the local, post-injection adverse events (AEs) in some subjects.

There has been a demand by physicians for an alternative to urinary products for treatment. Due to allergies to urinary products, or other personal reasons, subjects were not able or willing to be treated with proteins of human origin. This study allowed subjects to be treated with the recombinant human chorionic gonadotropin (r hCG) (free of urinary proteins), which otherwise would not be possible. The study sponsor used this opportunity to collect additional safety data on the new recombinant product, (Ovidrel, r-hCG).

DETAILED DESCRIPTION:
Approximately one in ten couples of reproductive age experiences infertility. Infertility may be caused by problems in men, in women or in both. A number of techniques can be used depending on the duration and type of infertility problems. The treatment of ovulation induction (OI) uses the help of exogenous gonadotrophins such as follicle stimulating hormone (FSH), luteinizing hormone (LH) and hCG in order to stimulate follicles and release oocytes for fertilization in the fallopian tubes.

Assisted reproductive technologies (ARTs), including in-vitro fertilization (IVF) and intra- cytoplasmic sperm injection (ICSI), increases the chances of success to obtain more than one embryo. In order to obtain more than one embryo, it is necessary to stimulate the growth and maturation of several follicles. Such a multiple follicular development is obtained by daily administration of a follicle stimulating hormone (r-hFSH, Gonal-F). When these follicles have reached a large enough size, the role of hCG is to achieve final oocyte maturation and initiation of follicular luteinization.

Serono International S.A. has developed a pharmaceutical preparation of human chorionic gonadotrophin (hCG) for clinical use through the application of recombinant DNA technology. The resulting product is choriogonadotrophin alpha, a pure recombinant human chorionic gonadotrophin (r-hCG). The corresponding drug product is marketed under the tradename Ovidrel. Ovidrel (choriogonadotrophin alpha for injection) has been approved in the United States, in the European Union and Australia.

OBJECTIVES The objective of this study was to collect safety information in order to confirm the already known profile of r- hCG (Ovidrel).

ELIGIBILITY:
Inclusion Criteria:

* Infertile women desiring a pregnancy
* Subjects whose baseline hormonal values were within normal ranges as per local practice
* Subjects who were willing and able to comply with the protocol for the duration of the study
* Subjects who had given written informed consent, prior to treatment, with the understanding that consent might be withdrawn at any time without prejudice

Exclusion Criteria:

* Subjects with clinically significant disease
* Subjects who were known to be infected by human immunodeficiency virus (HIV), Hepatitis B or C
* Subjects who had any medical condition, which in the judgment of the investigator, may interfere with the absorption, distribution, metabolism or excretion of study drug
* Subjects with severe endometriosis
* Subjects with abnormal, undiagnosed gynaecological bleeding
* Subjects who had any contra-indication to being pregnant or carrying a pregnancy to term
* Subjects who were pregnant or breast-feeding at the beginning of the cycle. Confirmation that the subject was not pregnant was to be established by a negative urine or serum pregnancy test in the 7 days prior to Study Day1
* Subjects with prior hypersensitivity to hCG preparations or one of their excipients
* Subjects with uncontrolled thyroid or adrenal dysfunction
* Subjects with uncontrolled organic intracranial lesion such as a pituitary tumour
* Subjects with ovarian cyst or enlargement of undetermined origin
* Subjects with sex hormone dependent tumors of the reproductive organs and breasts

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects desiring pregnancy who had been unable to conceive and been diagnosed by a physician who is familiar with infertility and its monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2003-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Pre-treatment screening within 6 weeks prior to beginning GnRH-agonist therapy or stimulation day 1 (S1) to post-treatment period (30 days of the last administration of the investigational product)
  Safety of Ovidrel was assessed through the recording, reporting and analysis of baseline medical conditions, adverse events, general physical examination, laboratory tests, and vital signs data.

CONTACTS AND LOCATIONS:
Overall Officials: Horia Ijacu, MD, Study Director — EMD Serono a division of EMD Canada Inc.